CLINICAL TRIAL: NCT01763320
Title: China Angioplasty & Stenting for Symptomatic Intracranial Severe Stenosis (CASSISS): a New, Prospective, Multi-center, Randomized Controlled Trial in China
Brief Title: China Angioplasty & Stenting for Symptomatic Intracranial Severe Stenosis
Acronym: CASSISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, jiaoliqun, MD.PhD, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XW125-S002
Record Dates: First submitted 2013-01-06; First posted 2013-01-08 (Estimated); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; intracranial stenting; vascular risk factor management
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracranial stenting group (Experimental): all the participants in this group will be performed with intracranial stenting
  Interventions: Procedure: Intracranial stenting group
- medical group (Active Comparator): all the participants in this group will be given medical therapy including aspirin 100mg + clopidogrel 75mg per day for 90 consecutive days and clopidogrel 75mg per day thereafter
  Interventions: Drug: medical group

INTERVENTIONS:
Procedure: Intracranial stenting group — all the participants in this group will be performed with intracranial stenting
  Arms: Intracranial stenting group
Drug: medical group — all the participants in this group will be given medical therapy including aspirin 100mg + clopidogrel 75mg per day for 90 consecutive days and clopidogrel 75mg per day thereafter
  Arms: medical group

SUMMARY:
Patients with symptomatic stenosis of intradural arteries are at high risk for subsequent stroke. Since the SAMMPRIS trial, stenting is no longer recommended as primary treatment, however, the results of this trial, its inclusion criteria and its center selection received significant criticism and did not appear to reflect our experience, neither regarding natural history, nor treatment complications rate. As ICAS is the most common cause for stroke in Asian countries, we are hereby proposing a refined prospective randomized multicenter study in an Asian population with strictly defined patient and participating center inclusion criteria.

The China Angioplasty & Stenting for Symptomatic Intracranial Severe Stenosis (CASSISS) trial, is an ongoing, government-funded, prospective, multicenter randomized trial. It recruits patients with recent TIA or stroke caused by 70-99% stenosis of a major intracranial artery. Patients with previous stroke related to perforator ischemia will not be included. Only high-volume center with a proven track record will enroll patients as determined by a lead-in phase. Patients will be randomized (1:1) to best medical therapy alone or medical therapy plus stenting. Primary endpoints are any stroke or death within 30 days after enrollment or after any revascularization procedure of the qualifying lesion during follow-up, or stroke in the territory of the symptomatic intracranial artery beyond 30 days The CASSISS trial will be conducted in 8 sites in China with core imaging lab review at a North American site and aims to have a sample size of 380 subjects (stenting, 190; medical therapy, 190). Recruitment is expected to be finished by Dec, 2016. Patients will be followed for at least three years. The trial is scheduled to complete in 2019. In the proposed trial, certain shortcomings of SAMMPRIS including patient and participating center selection will be addressed. The present manuscript outlines the rationale and design of the study. We estimate that this trial will allow for a critical reappraisal of the role of intracranial stenting for selected patients in high volume centers.

DETAILED DESCRIPTION:
Although SAMMPRIS trial has had an impact on the current treatment of intracranial atherosclerotic (ICAS), criticism regarding to its design were still raised and remained unsettled. In light of SAMMPRIS, medical therapy could not be good as it was; neither stenting for ICAD need to be abolished, but rather its role needs to be redefined by future prospective trials. Moreover, China is a developing country, and has the world's largest population. Since 2010, stroke has been the leading cause of death in China and confers a huge burden and effort on patients and health professionals. Compared with western countries, ICAS is the most common vascular lesion in patients with cerebro-vascular disease, and is an important cause of ischemic stroke and future recurrent events in China. However, its treatment strategy and long-term result has not been well determined. The health burden in China and ethnic difference of ICAS incidence as well as the willingness to continue clinical trials, support the need for ongoing CASSISS in China.

Pre-CASSISS registry trial:

A registration pilot trial was performed prior to CASSISS. It aimed to test the credentialing of interventionists and participating centers. From July 2013 to Mar 2014, 12 candidates were involved in a competitive registration study of recruiting 100 consecutive patients. The patients received stenting using Wingspan at each site. As for the candidate centers, the following aspects will be considered: stenting experiences, peri-operative complications, and the volume of stenting cases. Those met the following criteria were not involved into the subsequent randomization trial: 1) each center performed more than 5 procedures; 2) clinical results demonstrated the complication rates were more than 15% (stroke or death). At last, 4 sites were excluded and the remaining 8 were certified and invited for the final randomization trial.

ELIGIBILITY:
Inclusion criteria：

1. Eligible patients aged between 30-80 years; intracranial arterial stenosis related to the following non-atherosclerotic factors will be not be considered: arterial dissection, moya-moya disease; vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid pleocytosis; radiation-induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process, and suspected recanalized embolus;
2. Symptomatic ICAS: presented with TIA or stroke within the past 12 months attributed to 70%-99% stenosis of a major intracranial artery (internal carotid artery, MCA [M1], vertebral artery, or basilar artery);
3. Degree of stenosis: 70%-99%; stenosis degree must be confirmed by catheter angiography for enrollment in the trial;
4. There might be remote infarctions on MRI scan, which could be accounted by the occlusion of the terminal cortical branches or hemodynamic compromise (perforator occlusion excluded). Infarction due to perforators occlusion is defined as basal ganglia or brainstem/thalamus infarction related with MCA or BA stenosis;
5. Expected ability to deliver the stent to the lesion;
6. All the patients should be performed with stenting beyond a duration of 3 weeks from the latest ischemic symptom onset;
7. No recent infarctions identified on MRI (indicated as high signals on DWI series) upon enrollment;
8. No massive cerebral infarction (>1/2 MCA territory), intracranial hemorrhage, epidural or sub-dural hemorrhage, and intracranial brain tumor on CT or MRI scan;
9. mRS scale score of <=2;
10. Target vessel reference diameter must be measured to be 2.00 mm to 4.50 mm; target area of stenosis is <=14 mm in length;
11. No childbearing potential or has a negative pregnancy test within the past 1 week prior to study procedure; female patients had normal menses in the last 18 months;
12. Patient is willing and able to return for all follow-up visits required by the protocol;
13. Patients understand the purpose and requirements of the study and have signed informed consent form.

Exclusion criteria:

1. Refractory to general anesthesia; patients were not able to be overcome by pre-treatment with medical therapy.
2. Any condition that precludes proper angiographic assessment.
3. Tandem extracranial or intracranial stenosis (70%-99%) or occlusion that is proximal or distal to the target intracranial lesion.
4. Bilateral intracranial VA stenosis of 70%-99% and uncertainty about which lesion is symptomatic (e.g., if patient has pon, midbrain, temporal and occipital symptoms).
5. Presence of a previously placed intravascular stent or graft in the ipsilateral distribution within 30 days.
6. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform staged angioplasty followed by stenting of target lesion.
7. Severe vascular tortuosity or anatomy that would preclude the safe introduction of a guiding catheter, guiding sheath or stent placement.
8. Plan to perform concomitant angioplasty or stenting of an extracranial. vessel tandem to an ipsilateral intracranial stenosis.
9. Presence of intraluminal thrombus proximal to or at the target lesion.
10. Any aneurysm proximal to or distal to intracranial stenotic artery.
11. Intracranial tumors or any intracranial vascular malformations.
12. Computed tomographic or angiographic evidence of severe calcification at target lesion.
13. Thrombolytic therapy within 24 hours before enrollment.
14. Evolving stroke or progressive neurologic signs within 24 hours before enrollment.
15. Stroke of sufficient size (>5cm on CT or MRI) to place patient at risk of hemorrhagic transformation during the procedure; hemorrhagic transformation of an ischemic stroke within the past 15 days.
16. Previous spontaneous intracerebral (parenchymal) or other intracranial (subarachnoid, subdural, or epidural) hemorrhage within 30 days.
17. Untreated chronic subdural hematoma >5 mm in thickness.
18. Other cardiac sources of emboli such as left ventricular aneurysms, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcified aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, left atrial myxoma.
19. Myocardial infarction within previous 30 days.
20. Chronic atrial fibrillation; any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
21. Intolerance or allergic reaction to any of the medical therapy, including aspirin, clopidogrel, heparin, and local or general anesthetics.
22. History of life-threatening allergy to contrast medium. If not life-threatening and can be effectively pre-treated, patient can be enrolled at physicians' discretion.
23. Recent gastro-intestinal bleed that would interfere with anti-platelet therapy.
24. Active bleeding diathesis or coagulopathy; active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets count <125,000, hematocrit <30, Hgb <10 g/dl, uncorrected INR >1.5, bleeding time >1 minute beyond upper limit normal, or heparin-associated thrombocytopenia that increases the risk of bleeding, uncontrolled severe hypertension (systolic BP>180 mm hg or diastolic BP>115 mm hg), severe liver impairment (AST or ALT >3 times normal, cirrhosis), creatinine >265.2μmol/l (unless on dialysis)
25. Major surgery (including open femoral, aortic, or carotid surgery) within previous 30 days or planned in the next 90 days after enrollment.
26. Indication for warfarin or heparin beyond enrollment (note: exceptions allowed for use of systemic heparin during stenting procedure or subcutaneous heparin for deep venous thrombosis prophylaxis while hospitalized).
27. Inability to understand and cooperate with study procedures or sign informed consent
28. Severe dementia or psychiatric problems that prevent the patients from following an outpatient program reliably.
29. Pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study
30. Actively participating in another drug or device trial that has not completed the required protocol follow-up period.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
stroke or death within 30 days after enrollment, any stroke in the territory of the symptomatic intracranial artery beyond 30 days through 12 months | 12 months
  the number of participants who suffer from stroke or death within 30 days after enrollment, or any stroke in the territory of the symptomatic intracranial artery beyond 30 days through 12 months

SECONDARY OUTCOMES:
the number of participants who suffer from disabling stroke or death | within 3 years
  the number of participants who suffer from disabling stroke or death
the number of participants who suffer from stroke in the territory of qualifying artery | within 2 years
  the number of participants who suffer from stroke in the territory of qualifying artery
the number of participants who suffer from stroke in the territory of qualifying artery | within 3 years
  the number of participants who suffer from stroke in the territory of qualifying artery
the number of participants who survives in both groups | within 3 years
  the number of participants who survives in both groups
the number of participants who suffer from any stroke,TIA, or cardiovascular events | within 3 years
  the number of participants who suffer from any stroke,TIA, or cardiovascular events within 3 years

OTHER OUTCOMES:
the number of participants who suffer from stroke or death within 30 days after enrollment | within 30 days after enrollment
  the number of participants who suffer from stroke or death within 30 days after enrollment
the number of participants who suffer from any stroke, death in the territory of the symptomatic intracranial artery beyond 30 days through 12 months | beyond 30 days through 12 months
  the number of participants who suffer from any stroke, death in the territory of the symptomatic intracranial artery beyond 30 days through 12 months
the rate of restenosis (>50%) related to stenting within a follow-up of 36 months | within a follow-up of 36 months
  the rate of restenosis (>50%) related to stenting within a follow-up of 36 months
National Institutes of Health Stroke Scale (NIHSS) assessment within a follow-up of 36 months; | within a follow-up of 36 months
  National Institutes of Health Stroke Scale (NIHSS) assessment within a follow-up of 36 months;
modified Rankin Scale score (mRS) score within a follow-up of 36 months; | within a follow-up of 36 months
  modified Rankin Scale score (mRS) score (0-6) within a follow-up of 36 months;
Barthel index assessment within a follow-up of 36 months; | within a follow-up of 36 months
  Barthel index assessment within a follow-up of 36 months;
the compliance rate of the patients with regular medical therapy within a follow-up of 36 months; | within a follow-up of 36 months;
  the compliance rate of the patients with regular medical therapy within a follow-up of 36 months;

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, Principal Investigator — Xuanwu Hospital, Capital University of Medical Sciences, Beijing, China
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Beijing, China

REFERENCES:
- [Background] Feigin VL. Stroke epidemiology in the developing world. Lancet. 2005 Jun 25-Jul 1;365(9478):2160-1. doi: 10.1016/S0140-6736(05)66755-4. No abstract available. PMID 15978910
- [Result] Chimowitz MI, Lynn MJ, Derdeyn CP, Turan TN, Fiorella D, Lane BF, Janis LS, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Torbey MT, Zaidat OO, Rumboldt Z, Cloft HJ; SAMMPRIS Trial Investigators. Stenting versus aggressive medical therapy for intracranial arterial stenosis. N Engl J Med. 2011 Sep 15;365(11):993-1003. doi: 10.1056/NEJMoa1105335. Epub 2011 Sep 7. PMID 21899409
- [Result] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Result] Zaidat OO, Klucznik R, Alexander MJ, Chaloupka J, Lutsep H, Barnwell S, Mawad M, Lane B, Lynn MJ, Chimowitz M; NIH Multi-center Wingspan Intracranial Stent Registry Study Group. The NIH registry on use of the Wingspan stent for symptomatic 70-99% intracranial arterial stenosis. Neurology. 2008 Apr 22;70(17):1518-24. doi: 10.1212/01.wnl.0000306308.08229.a3. Epub 2008 Jan 30. PMID 18235078
- [Result] Fiorella D, Levy EI, Turk AS, Albuquerque FC, Niemann DB, Aagaard-Kienitz B, Hanel RA, Woo H, Rasmussen PA, Hopkins LN, Masaryk TJ, McDougall CG. US multicenter experience with the wingspan stent system for the treatment of intracranial atheromatous disease: periprocedural results. Stroke. 2007 Mar;38(3):881-7. doi: 10.1161/01.STR.0000257963.65728.e8. Epub 2007 Feb 8. PMID 17290030
- [Result] Derdeyn CP, Chimowitz MI, Lynn MJ, Fiorella D, Turan TN, Janis LS, Montgomery J, Nizam A, Lane BF, Lutsep HL, Barnwell SL, Waters MF, Hoh BL, Hourihane JM, Levy EI, Alexandrov AV, Harrigan MR, Chiu D, Klucznik RP, Clark JM, McDougall CG, Johnson MD, Pride GL Jr, Lynch JR, Zaidat OO, Rumboldt Z, Cloft HJ; Stenting and Aggressive Medical Management for Preventing Recurrent Stroke in Intracranial Stenosis Trial Investigators. Aggressive medical treatment with or without stenting in high-risk patients with intracranial artery stenosis (SAMMPRIS): the final results of a randomised trial. Lancet. 2014 Jan 25;383(9914):333-41. doi: 10.1016/S0140-6736(13)62038-3. Epub 2013 Oct 26. PMID 24168957
- [Derived] Gao P, He X, Wang H, Wang T, Wang D, Shi H, Li T, Zhao Z, Cai Y, Wu W, He W, Yu J, Zheng B, Feng X, Derdeyn CP, Dmytriw AA, Wu Y, Zhao G, Jiao L; CASSISS Trial Investigators. Stenting Versus Medical Therapy for Symptomatic Intracranial Artery Stenosis: Long-Term Follow-Up of a Randomized Trial. Stroke. 2025 May;56(5):1128-1137. doi: 10.1161/STROKEAHA.124.049602. Epub 2025 Mar 18. PMID 40099362
- [Derived] Wang T, Luo J, Li T, Almallouhi E, Gao P, Gong H, Zhang X, Wang J, Lu T, Yang Y, Yang R, Xing Z, Wang H, Derdeyn CP, Jiao L. Stenting versus medical treatment alone for symptomatic intracranial artery stenosis: a preplanned pooled individual patient data analysis. J Neurointerv Surg. 2025 Sep 12;17(10):1032-1039. doi: 10.1136/jnis-2024-022189. PMID 39147573
- [Derived] Gao P, Wang T, Wang D, Liebeskind DS, Shi H, Li T, Zhao Z, Cai Y, Wu W, He W, Yu J, Zheng B, Wang H, Wu Y, Dmytriw AA, Krings T, Derdeyn CP, Jiao L; CASSISS Trial Investigators. Effect of Stenting Plus Medical Therapy vs Medical Therapy Alone on Risk of Stroke and Death in Patients With Symptomatic Intracranial Stenosis: The CASSISS Randomized Clinical Trial. JAMA. 2022 Aug 9;328(6):534-542. doi: 10.1001/jama.2022.12000. PMID 35943472
- [Derived] Gao P, Wang D, Zhao Z, Cai Y, Li T, Shi H, Wu W, He W, Yin L, Huang S, Zhu F, Jiao L, Ji X, Qureshi AI, Ling F. Multicenter Prospective Trial of Stent Placement in Patients with Symptomatic High-Grade Intracranial Stenosis. AJNR Am J Neuroradiol. 2016 Jul;37(7):1275-80. doi: 10.3174/ajnr.A4698. Epub 2016 Feb 11. PMID 26869472